CLINICAL TRIAL: NCT00713752
Title: Establishing Normal Values for Neuropsychological Testing in HIV-negative Thais
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Responsible Party: Principal Investigator, Assoc.Prof.Jintanat Ananworanich, M.D., Assoc.Prof., SEARCH Research Foundation
Other Study IDs: SEARCH002
Record Dates: First submitted 2008-07-08; First posted 2008-07-11 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: HIV-negative
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to establish normal values for neuropsychological testing in HIV negative Thais stratified by age (1 decade) and education (no certificate or primary school certificate, less than high school certificate or vocational certificate, high school certificate or higher vocational certificate or diploma, Bachelor degree or higher.

DETAILED DESCRIPTION:
The Southeast Asia Research Collaboration with Hawaii (SEARCH) operates or collaborates on several neuroAIDS research protocols. To allow accurate interpretation of neuropsychological data, normative data that are obtained in a similar population are needed. Currently, there are limited such data available for this purpose.

The SEARCH 001 study evaluated the neurocognitive changes before and after highly active antiretroviral therapy in 30 HIV positive subjects and has also enrolled 230/300 proposed HIV-negative controls for this purpose. Normative data tables typically require many more individuals so that age and education strata can be established. We now propose to enroll up to 1000 HIV-seronegative individuals for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-69
2. Male or female
3. Negative HIV antibody at screening
4. Have the ability to understand the study and signed the informed consent form

Exclusion Criteria:

1. Head injury with loss of consciousness greater than 1 hour
2. Current or past illicit drug use or positive drug screen for amphetamine, methamphetamines, cocaine, marijuana, or narcotics
3. Severe illness within 30 days prior to entry
4. Current or recent fevers or meningeal signs.
5. History of pre-existing neurologic disease to include stroke, multiple sclerosis or autoimmune disease.
6. active major depression will be excluded as well - patients with past depression that is controlled and patients with or minor depressive symptoms will be allowed to enroll.
7. Known learning disability including dyslexia
8. Confusion or other signs and symptoms of metabolic encephalopathy or delirium
9. Focal neurological deficit on examination
10. Examining physician's concern that participant may not be able to complete visit requirements.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-negative Thais
Sampling Method: Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2008-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To establish normal values for neuropsychological testing in HIV negative Thais stratified by age (1 decade) and education | July 31, 2014

SECONDARY OUTCOMES:
To estimate the learning effect on these test at 6 months and 12 months. | July 31, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Victor - Valcour, M.D., Principal Investigator — University of Hawaii
Locations (1):
- SEARCH Thailand, Bangkok, Bangkok, Thailand